CLINICAL TRIAL: NCT00609765
Title: Phase II Study of Avastin, Fluorouracil, Doxorubicin and Streptozocin in Locally Advanced and Metastatic Pancreatic Endocrine Tumors
Brief Title: Avastin, Fluorouracil, Doxorubicin and Streptozocin in Locally Advanced and Metastatic Pancreatic Endocrine Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Development of new chemotherapy standard of care for treatment rendered the trial obsolete.
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14961; AVF3915s (Other: Genentech)
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Results first posted 2011-03-22 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2011-03

CONDITIONS: Pancreatic Cancer
Keywords: advanced; unresectable; metastatic; endocrine; tumors
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Bevacizumab; Fluorouracil; Doxorubicin; Streptozocin; Dexamethasone; Calcium Dobesilate; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Protocol Specified Chemotherapy (Experimental): Protocol Specified Chemotherapy Every 28 Days: Avastin, Fluorouracil, Doxorubicin, Streptozocin.
  Premedications: Dexamethasone, Ondansetron
  Interventions: Drug: Avastin; Drug: Fluorouracil; Drug: Doxorubicin; Drug: Streptozocin; Drug: Dexamethasone; Drug: Ondansetron

INTERVENTIONS:
Drug: Avastin — Every 28 Days: Avastin 5mg/kg iv days 1 and 15
  Other Names: bevacizumab
Drug: Fluorouracil — Every 28 Days: Fluorouracil 400mg/m^2 iv bolus daily days 1-5
  Other Names: Fluoroplex; 5-FU; Efudex
Drug: Doxorubicin — Every 28 Days: Doxorubicin 40mg/m^2 iv bolus day 1
  Other Names: Adriamycin®
Drug: Streptozocin — Every 28 Days: Streptozocin 400mg/m2 iv bolus daily days 1-5
  Other Names: Zanosar®
Drug: Dexamethasone — Premedication: Dexamethasone 20mg intravenously days 1-5
  Other Names: Decadron
Drug: Ondansetron — Premedication: Ondansetron 16mg intravenously days 1-5
  Other Names: Zofran

SUMMARY:
Open label, single-arm phase II study of avastin combined with fluorouracil, doxorubicin and streptozocin administered in 28-day cycles. Treatment will continue until progression of disease, or until withdrawal due to toxicity, or up to a maximum of 12 cycles (48 weeks). In order to reduce the risk of cardiac toxicity, doxorubicin will be administered for a maximum of 8 cycles. If disease has not progressed after 12 cycles of treatment, avastin monotherapy will continue until disease progression or withdrawal due to toxicity.

DETAILED DESCRIPTION:
Patients will need to come for 24 study visits in all. Most study visits will take about 2 hours. At some of these study visits, the doctor

* Will do a physical exam
* Will take blood for routine lab tests
* Will do a urinalysis
* Will administer study medication Some study visits may be longer because patient will have a CT scan or an MRI.

At patient's last visit, they will have a CT scan or MRI.

After treatment starts, patient will:

* Have their blood pressure monitored with every dose of Avastin® (about every 2 weeks).
* Have a history and physical with every chemotherapy cycle (about every 4 weeks).
* Have their blood taken for routine blood tests with every chemotherapy cycle (about every 4 weeks).
* Have a CT scan or MRI during every other cycle (about every 8 weeks).
* Have a MUGA scan during every 4 cycles (about 16 weeks).
* Have blood taken for tumor markers during every cycle only if their markers were high at baseline.
* Patients will receive study medication to treat their cancer:
* Fluorouracil on days 1 through 5 of each cycle through cycle 12
* Doxorubicin on day 1 of each cycle through cycle 8
* Streptozocin on days 1 through 5 of each cycle through cycle 12
* Avastin® on days 1 and 15 of each cycle through cycle 12

ELIGIBILITY:
Inclusion Criteria:

* Patients must have locally advanced (unresectable) or metastatic, well or moderately differentiated pancreatic endocrine tumors.
* Measurable disease on CT scan or MRI.
* Age ≥ 18 years and ≤ 80 years.
* Use of effective means of contraception (men and women) in subjects of child-bearing potential
* Adequate renal function (serum creatinine ≤1.5, urine protein:creatinine ratio <1.0 or urine dipstick for proteinuria < 2+ (patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1 g of protein in 24 hours to be eligible).
* Adequate hepatic function (bilirubin ≤2.0, AST and ALT ≤ 3x ULN.
* Adequate hematologic function (WBC ≥ 3,000, ANC ≥ 1500, platelets ≥ 100,000)

Exclusion Criteria:

* Prior therapy with fluorouracil, doxorubicin, streptozocin or avastin
* Ejection fraction on MUGA <50%
* ECOG performance status > 2
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored avastin cancer study
* Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* Unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Presence of central nervous system or brain metastases
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* Pregnant (positive pregnancy test) or lactating. Use of effective means of contraception (men and women) in subjects of child-bearing potential
* Proteinuria at screening as demonstrated by either

  * Urine protein: creatinine (UPC) ratio ≥ 1.0 at screening OR
  * Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
* Evidence of duodenal invasion on CT scan, MRI, or endoscopy
* Known hypersensitivity to any component of avastin
* Serious, non-healing wound, ulcer, or bone fracture
* Inability to comply with study and/or follow-up procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Kvols, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; Jonathan Strosberg, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy: Prospective, single arm, Phase II
Period: Overall Study
Arm/Group | Chemotherapy
Started | 1
Completed | 0
Not Completed | 1
Not completed — Study ended prior to 12 months | 1

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression Free Survival (PFS) at 12 Months
Description: We planned to calculate the One Year Progression Free Survival rate. The event for PFS analyses was the first occurrence of disease progression or death and patients who did not progress or died would be censored at the date of last tumor evaluation (e.g. one-year).
Time Frame: 12 months
Population: Per protocol at 12 months
Arm/Group | Chemotherapy
Number analyzed (Participants) | 0

2. Secondary Outcome: The Number of Participants With Radiographic Response
Description: Objective Radiographic Response Rate (ORR). We planned to calculate the sum of complete response (CR) and partial response (PR) in target lesions.
Time Frame: 2 years
Arm/Group | Chemotherapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Chemotherapy
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
This trial only enrolled one patient and was closed because of development of a new chemotherapy standard of care for treatment of this cancer which we felt rendered the trial obsolete. The trial was open for only 7 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No